CLINICAL TRIAL: NCT04525183
Title: REVITALIZE: A Telehealth Intervention for Women With Advanced Ovarian Cancer and PARP Inhibitor-Related Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AstraZeneca (Industry); National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Alexi A. Wright, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-285
Record Dates: First submitted 2020-08-10; First posted 2020-08-25 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Ovarian Cancer; Fatigue; Coping Behavior; Coping Skills
Keywords: Ovarian Cancer; Fatigue; Coping Behavior; Coping Skills
MeSH Terms: conditions — Ovarian Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Run In (Experimental): Recruit up to 5 patients who meet eligibility criteria to participate in the run-in period of the study
  * Participants will receive a 6-week Acceptance and Commitment Therapy (ACT) intervention (REVITALIZE).
  Interventions: Behavioral: REVITALIZE ACT Intervention
- Enhanced Usual Care (EUC) (Experimental): Participants randomized to EUC will receive educational materials developed by the National Comprehensive Cancer Network (NCCN) about fatigue and exercise during cancer treatment.
  Interventions: Behavioral: Enhanced Usual Care (EOC)
- REVITALIZE ACT Intervention (Experimental): Participants randomized to the REVITALIZE acceptance and commitment therapy (ACT) will receive 6 weekly sessions lasting approximately 60-75-minutes over a 6-8 week period, delivered face-to-face using iPads, computers or tablets, and a HIPAA-compliant platform (Zoom for Healthcare). If participants have difficulty connecting to the platform, telephone sessions are permitted.
  Interventions: Behavioral: REVITALIZE ACT Intervention

INTERVENTIONS:
Behavioral: Enhanced Usual Care (EOC) — Educational materials
  Arms: Enhanced Usual Care (EUC)
Behavioral: REVITALIZE ACT Intervention — Six 60-75 minute telehealth sessions approximately once a week for 6-8 weeks
  Arms: REVITALIZE ACT Intervention; Run In

SUMMARY:
This study is testing whether a 6 week skills-based telehealth intervention can help ovarian cancer patients experiencing PARP inhibitor-related fatigue reduce the impact of fatigue on their daily life and activities.

DETAILED DESCRIPTION:
This is a two-arm, multicenter pilot randomized controlled trial to compare the feasibility, acceptability, and preliminary efficacy of REVITALIZE, a 6-week Acceptance and Commitment Therapy (ACT) telehealth intervention vs. enhanced usual care (EUC) in fatigued patients with ovarian cancer on maintenance PARPi.

The intervention is called REVITALIZE, and it is a structured, skills-based intervention for providing support, knowledge, and skills for coping with fatigue. This type of intervention has been used in other studies to treat symptoms such as pain, migraines, or worry. This research is being done to develop this program at the Dana-Farber Cancer Institute and the University of Pennsylvania's Abramson Cancer Center, and to get patient feedback on the telehealth intervention to improve it for a future study. The study is also making a preliminary determinations as to whether REVITALIZE does improve psychological flexibility and fatigue-related interference and reduces fatigue, psychological distress, and fear of cancer recurrence, while improving overall quality of life (QOL).

The study will pre-pilot the REVITALIZE intervention in up to 5 patients at the Dana-Farber Cancer Institute (DFCI). This run-in phase serves to test and refine the newly developed 6-week ACT intervention in a smaller sample size prior to initiating the randomized control trial (RCT) portion of the study. After the ACT intervention has been tested and refined, the study will enroll and randomize 40 fatigued patients with advanced ovarian cancer on maintenance PARPi at Dana-Farber Cancer Institute and the Abramson Cancer Center at the University of Pennsylvania. Participants will be randomized to receive either a 6-week ACT intervention or enhanced usual care (educational materials). The study anticipates enrolling approximately 20 patients at each site, and 20 patients will be enrolled to each study arm. The ACT intervention will be delivered by masters' level psychologists at The University of Colorado Boulder.

It is expected participants will remain in the study for the duration of the intervention and follow-up assessments, which is approximately 3 months.

The Funding Organization for this study is the National Comprehensive Cancer Network (NCCN) and the Research Funding Provider is AstraZeneca.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years of age who have been diagnosed with epithelial ovarian, fallopian tube, or primary peritoneal carcinoma.
* Receiving PARPI inhibitors for ≥ 2 months.
* Able to read/speak English.
* Have an Eastern Oncology Group (ECOG) performance of 0-2.
* Report moderate-severe fatigue in the past week (average score ≥4 on a Fatigue Symptom Inventory scale of 0-10)

Exclusion Criteria:

* Patients with an untreated clinical condition or comorbid illness (e.g. anemia, hypothyroidism) that could explain their fatigue.
* Patients with chronic severe fatigue that pre-dates their use of PARPi.
* The following special populations will be excluded from this research:

  * Adults unable to consent
  * Individuals who are not yet adults (infants, children, teenagers)
  * Pregnant women
  * Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 49 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexi A Wright, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute; Joanna J Arch, PhD, Principal Investigator — University of Colorado, Boulder; Hanneke MD Poort, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Result] Wright AA, Poort H, Tavormina A, Schmiege SJ, Matulonis UA, Campos SM, Liu JF, Slivjak ET, Gilmour AL, Salinger JM, Haggerty AF, Arch JJ. Pilot randomized trial of an acceptance-based telehealth intervention for women with ovarian cancer and PARP inhibitor-related fatigue. Gynecol Oncol. 2023 Oct;177:165-172. doi: 10.1016/j.ygyno.2023.08.020. Epub 2023 Sep 13. PMID 37708581

RESULTS

PARTICIPANT FLOW:
Groups:
- Run-in Period: Tested and refined the REVITALIZE intervention in a sample of up to 5 patients with ovarian cancer who report fatigue associated with PARPi in a single-arm pre-pilot run-in phase of a 6-week ACT intervention (REVITALIZE).
Period: Overall Study
Arm/Group | Run-in Period | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention
Started | 4 | 23 | 21
Completed | 4 | 23 | 16
Not Completed | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Study non-compliance | 0 | 0 | 1
Not completed — Recurrent disease before starting on study | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (10.8) | 63.4 (9.5) | 62.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White/non-Hispanic | 20 | 20 | 40
  Race/Ethnicity: Asian/non-Hispanic | 2 | 1 | 3
  Race/Ethnicity: Other/non-Hispanic | 1 | 0 | 1
Education [Count of Participants; unit: Participants]
  High school or less | 2 | 2 | 4
  Some college | 6 | 3 | 9
  College or higher | 15 | 16 | 31
Employment [Count of Participants; unit: Participants]
  Full-time/part-time | 10 | 6 | 16
  Unemployed | 0 | 2 | 2
  Disabled | 2 | 1 | 3
  Retired | 11 | 11 | 22
  Other | 0 | 1 | 1
Relationship status [Count of Participants; unit: Participants]
  Married/Cohabitating | 17 | 14 | 31
  Single, never married | 4 | 1 | 5
  Divorced/separated | 2 | 4 | 6
  Widowed/other | 0 | 2 | 2
Ovarian cancer stage [Count of Participants; unit: Participants] — In order to classify the cancer stages for the participants in this study, the International Federation of Gynecology and Obstetrics (FIGO) system was used.
  STAGE I: Tumor confined to ovaries STAGE II: Tumor involves 1 or both ovaries with pelvic extension (below the pelvic brim) or primary peritoneal cancer Stage III: STAGE III: Tumor involves 1 or both ovaries with cytologically or histologically confirmed spread to the peritoneum outside the pelvis and/or metastasis to the retroperitoneal lymph nodes STAGE IV: Distant metastasis excluding peritoneal metastasis
  Participants
    Stage I-II | 4 | 4 | 8
    Stage III | 12 | 12 | 24
    Stage IV | 7 | 5 | 12
Germline mutation [Count of Participants; unit: Participants]
  Yes | 10 | 12 | 22
  No | 13 | 9 | 22
PARP inhibitor indication [Count of Participants; unit: Participants]
  Maintenance after first line | 8 | 12 | 20
  Maintenance for platinum-sensitive recurrence | 14 | 5 | 19
  Other | 1 | 4 | 5
Time on PARP inhibitor [Mean (Standard Deviation); unit: days] | 333.9 (302.9) | 453.2 (290.1) | 390.8 (299.5)
Time since diagnosis [Median (Inter-Quartile Range); unit: years] | 2.6 [1.1 to 2.9] | 2.2 [1.3 to 3.0] | 2.5 [2.3 to 2.7]

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Interference
Description: Changes in fatigue interference were measured using the validated 7-item interference scale of the Fatigue Symptom Inventory scale. Interference items assessed the degree to which fatigue interfered with general levels of activity, ability to bathe and dress, normal work activity, ability to concentrate, relations with others, enjoyment of life, and mood. Fatigue interference was scored on an 11-point scale, ranging from 0 (no interference) to 10 (extreme interference). Interference items were summed to obtain a total perceived interference score, with higher scores indicating greater fatigue interference.
Time Frame: Change from baseline to 4-, 8-, and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale (describing the units)
Arm/Group | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention
Number analyzed (Participants) | 23 | 21
score on a scale (describing the units)
  Baseline | 3.76 (2.04) | 3.52 (1.77)
  Week 4 | 2.80 (1.93) | 2.56 (1.25)
  Week 8 | 2.73 (2.10) | 2.43 (1.34)
  Week 12 | 2.96 (2.06) | 1.32 (1.14)

2. Primary Outcome: Fatigue Severity
Description: The Fatigue Symptom Inventory (FSI), is a 14-item self-report measure designed to assess the severity, frequency, and daily pattern of fatigue as well as its perceived interference with quality of life. Severity is measured on separate 11-point scales (0=not at all fatigued; 10=as fatigued as I could be) that assess most, least, and average fatigue in the past week as well as current fatigue. Frequency is measured as the number of days in the past week (0-7) that respondents felt fatigued as well as the extent of each day on average they felt fatigued (0=none of the day; 10=the entire day). Perceived interference is measured on separate 11-point scales (0=no interference; 10=extreme interference) that assess the degree to which fatigue in the past week was judged to interfere with general level of activity, ability to bathe and dress, normal work activity, ability to concentrate, relations with others, enjoyment of life, and mood. Higher FSI scores are associated with worse outcomes.
Time Frame: Change from baseline to 4-, 8-, and 12-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention
Number analyzed (Participants) | 23 | 21
units on a scale
  Baseline | 5.03 (1.21) | 5.05 (0.91)
  Week 4 | 3.88 (1.55) | 4.36 (1.43)
  Week 8 | 4.06 (1.75) | 4.16 (1.25)
  Week 12 | 4.22 (1.81) | 3.33 (1.35)

3. Primary Outcome: Current Fatigue
Description: as for outcome 2
Time Frame: Change from baseline to 4-, 8-, and 12-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention
Number analyzed (Participants) | 23 | 21
units on a scale
  Baseline | 4.52 (2.31) | 4.52 (1.57)
  Week 4 | 3.48 (2.23) | 4.33 (2.32)
  Week 8 | 4.04 (2.50) | 4.00 (2.00)
  Week 12 | 4.17 (2.67) | 2.73 (1.62)

4. Secondary Outcome: Emotional Distress: Anxiety Symptoms
Description: Emotional distress was assessed using the Generalized Anxiety Disorder 7-Item (GAD-7), which is a reliable and validated self-report measure to assess anxiety symptoms. For the GAD-7, respondents rated how often they have been bothered by 7 anxiety symptoms over the past 2 weeks using the following scale: 0 = Not at all; 1 = Several Days; 2 = Over half the days; and 3 = Nearly every day. Respondents also answer a question to assess the duration of their anxiety symptoms. The scale is scored 0-21, where 0-4 is minimal anxiety, 5-9 is mild anxiety, 10-14 is moderate anxiety, and scores >15 is severe anxiety. Using a cut-off of 8 the GAD-7 has a sensitivity of 92% and specificity of 76% for diagnosis generalized anxiety disorder.
Time Frame: Change from baseline to 4-, 8-, and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale (describing the units)
Arm/Group | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention
Number analyzed (Participants) | 23 | 21
score on a scale (describing the units)
  Baseline | 5.84 (4.88) | 5.85 (4.75)
  Week 4 | 5.51 (4.50) | 4.12 (2.71)
  Week 8 | 6.14 (5.34) | 3.94 (3.36)
  Week 12 | 5.32 (4.91) | 2.83 (1.76)

5. Secondary Outcome: Fear of Cancer Recurrence
Description: Fear of cancer recurrence will be measured using the 42-item Fear of Cancer Recurrence Inventory (FCRI). This survey has been validated across diverse cancer populations, has strong psychometric qualities, and is the most comprehensive multidimensional scale of FCR available.[36, 37] Items are scored on a Likert scale ranging from 0 ("not at all" or "never") to 4 ("a great deal or "all the time"). Higher scores indicate higher FCR. The FCRI is both internally consistent (Cronbach's α=0.75 to 0.91 across subscales) and stable over a two-week interval (ρ = 0.58 to 0.83 across subscales). It also has convergent validity with other standardized measures of FCR (ρ = 0.66 to 0.77) and discriminant validity with QOL amongst a large sample (n = 600) of Canadian cancer patients with varying tumor types.
Time Frame: Change from baseline to 4-, 8-, and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale (describing the units)
Arm/Group | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention
Number analyzed (Participants) | 23 | 21
score on a scale (describing the units)
  Baseline | 88.2 (27.2) | 83.6 (20.2)
  Week 4 | 81.5 (27.7) | 72.9 (19.8)
  Week 8 | 81.0 (30.4) | 74.0 (23.0)
  Week 12 | 78.6 (26.1) | 66.9 (23.1)

6. Secondary Outcome: Participant Quality of Life
Description: Participants' quality of life (QOL) was assessed with the Functional Assessment of Cancer Therapy-Ovarian Cancer (FACT-O), which has demonstrated internal consistency, reliability, and validity. This measure is composed of the Functional Assessment of Cancer Therapy-General scale, with an ovarian cancer-specific subscale (OCS) included. The measure is divided into five primary QOL domains: physical well-being (7-items, scored 0-28), social/family well-being (7-items, scored 0-28), emotional well-being (6-items, scored 0-24), functional well-being (7-items, scored 0-28), and additional concerns (OCS subscale, 12-items, scored 0-44). Participants rated each QOL domain item based on the past 7 days as: 0) Not at all; 1) A little bit; 2) Somewhat, 3) Quite a bit, and 4) Very much. Subscales can be analyzed separately or aggregated to produce a total score which is scored 0-152 with higher scores signifying better quality of life.
Time Frame: Change from baseline to 4-, 8-, and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale (describing the units)
Arm/Group | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention
Number analyzed (Participants) | 23 | 21
score on a scale (describing the units)
  Baseline | 60.39 (12.70) | 60.76 (11.43)
  Week 4 | 64.09 (14.10) | 64.15 (12.05)
  Week 8 | 63.30 (15.01) | 66.37 (12.09)
  Week 12 | 61.63 (14.60) | 69.81 (11.01)

7. Secondary Outcome: Emotional Distress: Depressive Symptoms
Description: We assessed emotional distress with the 8-item Patient Health Questionnaire (PHQ-8), which is a reliable and validated self-report measure to assess depressive symptoms. For the PHQ-8, respondents rated how often they have been bothered by 8 symptoms of depression over the past 2 weeks using the following scale: 0 = Not at all; 1 = Several Days; 2 = Over half the days; and 3 = Nearly every day. The scale is totaled (range 0-24) where total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Time Frame: Change from baseline to 4-weeks, 8-weeks, and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale (describing the units)
Arm/Group | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention
Number analyzed (Participants) | 23 | 21
score on a scale (describing the units)
  Baseline | 7.14 (4.05) | 7.14 (3.88)
  4 weeks | 6.17 (4.66) | 4.60 (2.41)
  8 weeks | 6.13 (4.24) | 4.27 (2.02)
  12 weeks | 6.13 (4.24) | 3.98 (2.12)

8. Other Pre Specified Outcome: Adherence
Description: We examined the number of participants who required reductions in the dose of their PARP inhibitor during the trial.
Time Frame: Change from baseline to 12-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention
Number analyzed (Participants) | 21 | 15
Participants
  Dose reduction | 4 | 1
  No dose reduction | 17 | 14

9. Other Pre Specified Outcome: Catastrophizing
Description: We assessed participants tendency to catastrophize about their fatigue using the Fatigue Catastrophizing Survey (FCS). Patients rate each question on a 5-point scale (1=never true to 5=all of the time) to indicate how often each item is true for them when they've experienced fatigue. The scale is scored by totaling the 10 items (range 10-50, where higher scores mean more severe fatigue catastrophizing). In prior research, more catastrophizing (as indicated by higher scores on the FCS) were associated with significantly greater fatigue.
Time Frame: Change from baseline to 4-, 8-, and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale (describing the units)
Arm/Group | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention
Number analyzed (Participants) | 23 | 21
score on a scale (describing the units)
  Baseline | 19.07 (8.86) | 17.58 (7.13)
  Week 4 | 17.35 (5.62) | 15.09 (4.01)
  Week 8 | 17.71 (6.76) | 15.33 (4.62)
  Week 12 | 17.57 (6.11) | 13.20 (2.81)

10. Other Pre Specified Outcome: Fatigue Self-Efficacy
Description: Self-efficacy concerning fatigue (i.e. the belief in one's capabilities to execute behaviors) was measured with the 7-item Self-Efficacy Scale (SES28). Items are scored on a 4-point Likert scale, and total scores range from 4 to 28. Higher scores indicate a greater sense of control over fatigue.
Time Frame: Change from baseline to 4-, 8-, and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale (describing the units)
Arm/Group | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention
Number analyzed (Participants) | 23 | 21
score on a scale (describing the units)
  Baseline | 19.48 (3.22) | 19.90 (2.19)
  Week 4 | 20.39 (3.2) | 21.73 (2.66)
  Week 8 | 19.74 (3.26) | 21.93 (3.13)
  Week 12 | 20.09 (3.50) | 22.27 (2.84)

11. Other Pre Specified Outcome: Psychological Flexibility
Description: We will measure changes in psychological flexibility (ACT processes) using the Acceptance and Action Cancer questionnaire, which is a 18-item measure adapted from the widely validated AAQ-II and diabetes-adapted AAQ towards cancer specific items. Numerous adaptations of the AAQ towards specific clinical targets have been shown to produce valid measures that mediate ACT outcomes for the specific population. The scale is scored by totaling the individual items (scale: 18-126). Lower scores reflect more psychological flexibility.
Time Frame: Change from baseline to 4-, 8-, and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale (describing the units)
Arm/Group | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention
Number analyzed (Participants) | 23 | 21
score on a scale (describing the units)
  Baseline | 51.11 (18.23) | 48.26 (16.06)
  4 weeks | 49.25 (18.11) | 41.56 (16.62)
  8 weeks | 47.64 (20.68) | 43.12 (16.30)
  12 weeks | 49.08 (18.26) | 36.31 (10.75)

12. Other Pre Specified Outcome: Experiential Avoidance
Description: Experiential avoidance will be measured using the Brief Multidimensional Experiential Avoidance Questionnaire (BEAQ) which only includes 15-items and covers all dimensions of experiential avoidance, including: behavioral avoidance, distress aversion, procrastination, distraction and suppression, repression and denial, and distress endurance. The scale is scored by totaling individual items (range 15-90), where higher scores reflect more avoidance. This measure is internally consistent and has been broadly associated with psychopathology and quality of life.
Time Frame: Change from baseline to 4-, 8-, and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale (describing the units)
Arm/Group | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention
Number analyzed (Participants) | 23 | 21
score on a scale (describing the units)
  Baseline | 40.17 (9.57) | 40.90 (13.43)
  4 weeks | 40.26 (11.43) | 35.80 (11.49)
  8 weeks | 39.64 (9.62) | 36.08 (12.07)
  12 weeks | 41.41 (11.61) | 33.40 (12.39)

13. Other Pre Specified Outcome: Value: Progress
Description: We will use the 10-item Valuing Questionnaire (VQ) to assess personal values enactment during the past two weeks. Respondents rate on a 6 point scale (0 "not at all true" to 6 "completely true") how often each item was true for them during the past two weeks and evaluate using a two-factor scale; the Progress scale and Obstruction scale. The scale is scored by totaling 5 individual items (scored 0-30), where higher progress scores are associated with positive affect, satisfaction with life, purpose in life and mastery and self-acceptance.
Time Frame: Change from baseline to 4-, 8-, and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale (describing the units)
Arm/Group | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention
Number analyzed (Participants) | 23 | 21
score on a scale (describing the units)
  Baseline | 22.91 (5.14) | 23.93 (4.61)
  4 weeks | 20.78 (7.15) | 23.28 (5.97)
  8 weeks | 22.67 (6.26) | 26.00 (4.00)
  12 weeks | 23.00 (5.16) | 25.27 (5.15)

14. Other Pre Specified Outcome: Valuing: Obstruction
Description: We will use the 10-item Valuing Questionnaire (VQ) to assess personal values enactment during the past two weeks. Respondents rate on a 6 point scale (0 "not at all true" to 6 "completely true") how often each item was true for them during the past two weeks and evaluate using a two-factor scale; the Progress scale and Obstruction scale. The VQ Obstruction subscale is scored by totaling the sum of 5 items (scored 0-30) Higher VQ Obstruction scores are associated with more depressive symptoms and negative affect.
Time Frame: Change from baseline to 4-, 8-, and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale (describing the units)
Arm/Group | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention
Number analyzed (Participants) | 23 | 21
score on a scale (describing the units)
  Baseline | 11.72 (5.03) | 11.93 (4.75)
  4 weeks | 11.26 (5.45) | 10.47 (4.37)
  8 weeks | 10.35 (5.12) | 8.93 (4.43)
  12 weeks | 12.13 (5.47) | 9.87 (4.49)

ADVERSE EVENTS:
Time Frame: Adverse events were collected on an ongoing basis throughout the course of the study, Day 1-90
Arm/Group | Enhanced Usual Care (EUC) | REVITALIZE ACT Intervention
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 0/23 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT04525183/Prot_SAP_000.pdf